CLINICAL TRIAL: NCT02303301
Title: Changes in the Oropharyngeal Flora in Hospitalised Patients
Brief Title: Changes of Oropharyngeal Flora
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Probi AB (Industry)
Responsible Party: Principal Investigator, Bengt Klarin, MD Consultant, Region Skane
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: ProOro
Record Dates: First submitted 2014-11-25; First posted 2014-11-27 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Pharyngeal Bacterial Colonization; Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Probiotics; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotics (Active Comparator): Patients gurgle twice a day with a suspension of two probiotic strains of bacteria- Contains also a filling material - maltodextrin
  Interventions: Dietary Supplement: Probiotics
- Control (Placebo Comparator): Patients gurgle twice a day with a suspension of the filling material - maltodextrin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics — Cultures from the oropharynx
  Other Names: ProViva (Lactobacillus plantarum 299v)
  Arms: Probiotics
Dietary Supplement: Placebo — Cultures from the oropharynx
  Other Names: Maltodextrin
  Arms: Control

SUMMARY:
Hospitalised patients have in contrast to healthy people enteric pathogenic bacteria in their oropharynx Increased risk of pneumonia due to the pathogens in the oropharynx Probiotics can reduce such bacteria in intubated critically ill patients This study will use two strain of probiotic bacteria for half of the patients and a placebo for the rest Active arm gurgles with a suspension twice a day Cultures at inclusion and at set time intervals The results of cultures from the two groups will be compared as will the use of antibiotics

DETAILED DESCRIPTION:
When patients are admitted to hospital some of them are already colonized in the oropharynx with pathogens that are normally found as commensal or possible pathogens in the gastrointestinal tract. This is probably a consequence of the illness that is the cause of their hospital admission.

Most patients admitted to hospital are elderly. Those patients often have their natural functions down regulated including their ability to secure their airway from aspiration. Acute illness whether you are old or young leads to changes in the intestinal microbiological flora. Bacteria normally found in the colon or distal ileum frequently appear in the stomach and more alarming in the oropharynx. Weakened by the illness, acute or chronic, there is an increased risk of aspiration and when there are pathogenic bacteria in the oropharynx, aspiration is likely to induce pneumonia - health related pneumonia.

For intubated ICU patients we have demonstrated a reduction of colonization with enteric bacteria by applying probiotics in the mouth.

After a screening period to find out what groups of patients that are most vulnerable, we will in a randomised way give probiotics to half of the included patients and to the other patients only the filling material (maltodextrin).

With this procedure our aim is to show a reduction of pathogens in the oropharynx and as a secondary outcome we hope to see a reduction of pneumonia.

Samples for microbiological analysis will be taken during the first day of admission to hospital and then at specified intervals.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to hospital
* Anticipated length of hospital stay 3 days or more

Exclusion Criteria:

* Immune insufficiency
* Prior participation in the study
* Not being able to understand study information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2014-10; Primary Completion 2019-03 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
New appearing pathogenic bacteria in the oropharynx | During hospital stay, Average 7 days
  Oropharyngeal cultures taken at admission and at specified days thereafter in all patients Results from Clin Microbiology assessed and all relevant findings will be treated according to patterns of antibiotic resistance

SECONDARY OUTCOMES:
Pneumonia | During hospital stay, Average 7 days
  Appearing health care related pneumonia. Treating physicians at the wards follow the patients condition and progress. Ward physicians prescribes antibiotics and chest x-rays on clinical grounds
Length of hospital stay | During hospital stay, Average 7 days
  Hospital stay , Days

CONTACTS AND LOCATIONS:
Overall Officials: Bengt Klarin, MD, PhD, Principal Investigator — Lund University Hospital
Locations (1):
- Lund University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Study results will be published as a scientific article

REFERENCES:
- [Background] Johanson WG, Pierce AK, Sanford JP. Changing pharyngeal bacterial flora of hospitalized patients. Emergence of gram-negative bacilli. N Engl J Med. 1969 Nov 20;281(21):1137-40. doi: 10.1056/NEJM196911202812101. No abstract available. PMID 4899868
- [Result] Klarin B, Molin G, Jeppsson B, Larsson A. Use of the probiotic Lactobacillus plantarum 299 to reduce pathogenic bacteria in the oropharynx of intubated patients: a randomised controlled open pilot study. Crit Care. 2008;12(6):R136. doi: 10.1186/cc7109. Epub 2008 Nov 6. PMID 18990201
- [Derived] Tranberg A, Klarin B, Johansson J, Pahlman LI. Efficacy of Lactiplantibacillus plantarum 299 and 299v against nosocomial oropharyngeal pathogens in vitro and as an oral prophylactic treatment in a randomized, controlled clinical trial. Microbiologyopen. 2021 Jan;10(1):e1151. doi: 10.1002/mbo3.1151. Epub 2020 Dec 22. PMID 33350604
- See also: Producers of the study products — http://www.probi.se